CLINICAL TRIAL: NCT04904120
Title: A Phase 1 Cross-over Biodistribution Study of [203Pb]VMT01 for Single Photon Emission Computed Tomography (SPECT) Imaging and [68Ga]VMT02 for Positron Emission Tomography (PET) Imaging of Stage IV Metastatic Melanoma
Brief Title: Targeted Imaging of Melanoma for Alpha-Particle Radiotherapy
Acronym: TIMAR1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Perspective Therapeutics (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: TIMAR1
Record Dates: First submitted 2021-05-03; First posted 2021-05-27 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2022-06

CONDITIONS: Melanoma (Skin); Melanoma Stage IV; Melanoma, Uveal; Melanoma, Mucosal
Keywords: Melanoma; Theranostic; Radiopharmaceutical; Radiotherapy; Alpha-Particle; Diagnostic; Metastatic; Single Photon Emission Computed Tomography (SPECT); Positron Emission Tomography (PET); Melanocortin Receptor Sub-type 1 (MC1R); VMT01; VMT02; Pb-203; Ga-68; Cancer; Immunohistochemistry (IHC)
MeSH Terms: conditions — Melanoma; Uveal Melanoma; Disease; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Archived tumor tissue will be tested for expression of the imaging target, melanocortin receptor sub-type 1 (MC1R). The qualified researcher who tests the sample, and the independent pathologist who reviews the results, will be blinded to a participant's identifying information and imaging results. Evaluators will not have access to the medical record.
  A pool of three qualified readers will evaluate study images (PET/CT and SPECT/CT). Images and medical information given to the readers will not include a participant's identifying information. The reader pool will not know the sequence of imaging for a participant or have access to the medical record.
  An independent medical physicist will validate imaging results and measurements of radiation absorbed and excreted by the participant's body. The physicist will be blinded to participant identifiers and demographics, as well as the sequence of imaging for a participant. The physicist will not have access to the medical record.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- [203Pb]VMT01 first (Active Comparator): Participants randomized to this arm will receive imaging agent [203Pb]VMT01 and undergo SPECT/CT imaging first. Later, participants in this arm will receive [68Ga]VMT02 and undergo PET/CT imaging.
  Interventions: Drug: [203Pb]VMT01; Drug: [68Ga]VMT02
- [68Ga]VMT02 first (Active Comparator): Participants randomized to this arm will receive imaging agent [68Ga]VMT02 and undergo PET/CT imaging first. Later, participants in this arm will receive [203Pb]VMT01 and undergo SPECT/CT imaging.
  Interventions: Drug: [203Pb]VMT01; Drug: [68Ga]VMT02

INTERVENTIONS:
Drug: [203Pb]VMT01 — Diagnostic imaging radiopharmaceutical; by intravenous infusion
Drug: [68Ga]VMT02 — Diagnostic imaging radiopharmaceutical; by intravenous infusion

SUMMARY:
The study hypothesis is that new imaging agents [203Pb]VMT01 and [68Ga]VMT02 can be safely used in humans without independent biological effect and can be used to image melanoma tumors expressing the melanocortin sub-type 1 receptor (MC1R) by SPECT/CT and PET/CT imaging modalities respectively.

DETAILED DESCRIPTION:
This is a first-in-human study evaluating the suitability of [203Pb]VMT01 for SPECT/CT imaging and [68Ga]VMT02 for PET/CT imaging of MC1R-expressing metastatic melanoma. Study results will provide foundational data to develop imaging and dosing for future therapeutic trials of [212Pb]VMT01 for the treatment of metastatic melanoma.

The study will be a cross-over study with the participants serving as their own comparator. Participants with positive FDG-PET scans for stage IV (or inoperable stage III) metastatic melanoma will undergo SPECT/CT scans utilizing [203Pb]VMT01 followed a few weeks later by PET/CT scans utilizing [68Ga]VMT02, or vice versa. The order of the imaging agents will be randomly assigned.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Stage IV metastatic melanoma, or inoperable Stage III equivalent
2. Baseline fluorodeoxyglucose (FDG)-PET scan available from within 30 days prior to date of enrollment
3. Blood counts and metabolic results within protocol limits within 14 days prior to enrollment
4. Ability to lie flat and still for a minimum of two hours for imaging
5. Male and female participants with reproductive potential must agree to use highly effective contraception in preparation of the study, during the study, and for 4 weeks following the last dose of an investigative imaging agent
6. Documented life expectancy of at least 3 months

Exclusion Criteria:

1. Active secondary malignancy
2. Prior treatment (for any reason) with radioactive nuclides; imaging tracers are acceptable
3. Pregnancy or breast feeding a child
4. Uncontrolled infection
5. Treatment with another investigational drug within 30 days prior to enrollment date
6. Any treatment with BRAF inhibitors since the baseline FDG-PET scan or plans for such treatment during the study
7. Kidney function not within protocol limits
8. BMI>40 kg/m2
9. History of a condition resulting in anaphylaxis or angioedema

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Study Imaging Agent-Associated Adverse Events (AE) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. | Visit 1 (Day 1) through Visit 5 (approximately Day 60 but could extend up to Day 108); ongoing Serious Adverse Events (SAE) will be followed for no longer than Day 65 or 30 days from the date of the SAE report (whichever is later).
  Adverse Events (AEs) will be assessed for severity according to CTCAE v5.0 and for relatedness to each of the investigative imaging agents ([203Pb]VMT01 and [68Ga]VMT02). Assessments attributed as possibly, probably, or definitely related to the imaging agent will be considered related.
Biodistribution of [68Ga]VMT02 | 12 hours
  Biodistribution will be calculated by utilizing PET/CT scans.
Biodistribution of [203Pb]VMT01 | 24 hours
  Biodistribution will be calculated by utilizing SPECT/CT scans.
Peak Plasma Concentration (Cmax) of [203Pb]VMT01 | 24 hours
  Cmax will be determined by blood sampling and direct radioactivity measurements.
Area Under the Plasma Concentration Versus Time Curve (AUC) for [203Pb]VMT01 | 24 hours
  AUC will be determined by blood sampling and direct radioactivity measurements.
Renal Excretion of [203Pb]VMT01 | 24 hours
  Renal excretion will be determined by urine sampling and direct radioactivity measurements.
Modeling of [203Pb]VMT01 Dosimetry | 24 hours
  Dosimetry will be modeled by utilizing the SPECT/CT scans.

SECONDARY OUTCOMES:
MC1R Expression Correlation Between Archived Tumor Tissue and Study Imaging | Historical tissue sample (collected <365 days before study enrollment) compared to Visit 1 (Day 1) and Visit 3 (Day 21-34) imaging
  Archived (previously collected) tumor tissue will be tested for MC1R expression and compared to study images obtained using MC1R targeted imaging agents, [203Pb]VMT01 and [68Ga]VMT02. The data will be assessed for an association between positive tissue and positive images.
Cancer Site Correlation Between Standard of Care Imaging Compared to Study Imaging | Historical imaging information compared to Visit 1 (Day 1) and Visit 3 (Day 21-34) imaging
  Sites of cancer detected previously by imaging will be compared to the presence or absence of positive imaging scans with the study agents, [203Pb]VMT01 and [68Ga]VMT02.
Dosimetry will be Calculated for each Study Imaging Agent by Measuring the Cumulative Absorbed Dose of Radiation to the Participant's Individual Organs and Tumors | Visit 1 (Day 1) and Visit 3 (Day 21-34) imaging
  For a given participant, dosimetry calculations will be compared between the two imaging agents with respect to cumulative absorbed dose of radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Frances L Johnson, MD, Principal Investigator — Perspective Therapeutics; Geoffrey B Johnson, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data (IPD) that underlies results in a peer-reviewed scientific publication will be shared.